CLINICAL TRIAL: NCT01929850
Title: Bariatric Surgery Plus Weight Watchers vs. Weight Watchers in Underserved Minorities: Randomized Controlled Cross-over Trial
Brief Title: Laparoscopic Sleeve Gastrectomy Plus Weight Watchers vs. Weight Watchers Alone in Underserved Minority Women
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Scientific/feasibility approval required prior to IRB review
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12-10409
Record Dates: First submitted 2013-08-15; First posted 2013-08-28 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Active Comparator): Sleeve gastrectomy laparoscopic surgery plus Weight Watchers for morbidly obese patients
  Interventions: Procedure: Laparscopic Sleeve Gastrectomy; Behavioral: Weight Watchers Program
- Control (Other): Weight Watchers Program for morbidly obese patients.
  Interventions: Behavioral: Weight Watchers Program

INTERVENTIONS:
Procedure: Laparscopic Sleeve Gastrectomy — The laparoscopic sleeve gastrectomy involves the placement of 5 trocars. A leak check may be performed at the same time by insufflating with a gastroscope with the remnant gastric section submerged in irrigation fluid and by infusing sterile methylene blue through a nasogastric tube. The staple line may be oversewn (3-0 Vicryl, Ethicon), only along the bleeding and leakage areas, or areas with the potential for such complications. A nasogastric decompression tube placed to monitor bleeding and an intraperitoneal drain was placed under an anastomotic stoma.
  Arms: Surgery
Behavioral: Weight Watchers Program — Intensive medically supervised nutritional and exercise therapy
  Other Names: Weight Watchers 360

SUMMARY:
Obesity is a costly multi-etiology world disease of fat storage. Morbid obesity is defines as greater than 100 pounds overweight and/or greater than 200 % of ideal body weight. Chronic underemployment, poor housing, child abuse, limited education, stress and anxiety are all associated with maternal morbid obesity. These latter conditions leave many patients in a state of economic, social and emotional poverty with need for life-long welfare support. For patients with true morbid obesity a standard surgical procedure is currently the procedure of choice especially among patients who fail standard medical intervention. The major procedures performed for morbid obesity include the Roux-en-Y gastric bypass, sleeve gastrectomy and laparoscopic band procedure. The sleeve gastrectomy is purely a restrictive procedure without malabsorptive components which involves one single staple line and can be performed laparoscopically in less than one hour. While these surgical procedures are recognized as "standard" procedures for patient who have failed medical treatment and are "covered" by most health plans, access to these procedures is limited for the medically underserved, rural, poor or underrepresented minorities since national, state and municipal health plans either provide minimal coverage or no coverage at all for surgery for morbid obesity. Reimbursement to providers offering these procedures is minimal and thus access to bariatric surgery is unlikely within a timely fashion.

DETAILED DESCRIPTION:
Obesity is a costly multi-etiology world disease of fat storage. Morbid obesity is defined as greater than 100 pounds overweight and/or greater than 200 % of ideal body weight. A commonly used measure of body mass is the Body Mass Index, BMI, which is the weight in kilograms divided by the body surface area in meters squared (kg/m²). A BMI greater than or equal to 40 is defined as morbid obesity. Morbid obesity is associated with an extraordinarily high increased risk of mortality principally from cardiovascular and cerebrovascular diseases. Morbidly obese patients routinely develop early hypertension, hypercholesterolemia, and diabetes mellitus. Currently, we estimate that approximately 15% of the adult U.S. population is morbidly obese. Morbid obesity is certainly not solely a disease of the economically advantaged. In developed countries where calories are readily available and relatively inexpensive, morbid obesity is disproportionately noted in culturally and economically disadvantaged people. Most disturbing, morbid obesity is especially prevalent among lower socioeconomic women between the ages of 21-40 years, when such women are bearing and rearing children. Morbid obesity for this patient population is clearly associated with the "Metabolic Syndrome" including such documented medical conditions such as diabetes, hypertension, sleep apnea, hypercholesterolemia and ultimately early onset heart disease and chronic lung disease. In addition, chronic underemployment, poor housing, child abuse, limited education, stress and anxiety are all associated with maternal morbid obesity. These latter conditions leave many patients in a state of economic, social and emotional poverty with need for life-long welfare support. The impact on the next generation reared by these morbidly obese underserved minority patients is likely to be dire.

Currently the major treatment programs available for morbid obesity including supervised dietary programs, pre-planned meals, positive reinforcement, and even pharmacological therapies are costly and have a very low permanent success rate. For patients with true morbid obesity a standard surgical procedure is currently the procedure of choice especially among patients who fail standard medical intervention.

One of the best known international programs is Weight Watchers International. Recent studies have documented weight loss of greater to or equal to 5 kg over a 12 month period.

Weight Watchers is an international company based in the United States that offers various products and services to assist weight loss and maintenance. It was founded in 1963 and operates in about 30 countries world-wide. The Weight Watcher's philosophy is to use a science-driven approach to help participants lose weight by forming helpful habits, eating smarter, getting more exercise and providing support. Weight Watchers uses the PointPlus System. This system is a calculation based on dietary protein, carbohydrates, fat and fiber. The weekly program focuses on assisting members in creating a caloric deficit to lose weight. The Weight Watchers Program is designed to result in a weight loss of ½ to 2 pounds per week. Members of Weight Watchers will be expected to go to hourly weekly meetings for selected topic discussions and to "weigh-in". Membership in the Weight Watchers Program includes not only weekly meetings, but also access to the Weight Watchers online, access to the Weight Watchers eTools and access to the Weight Watchers mobile applications.

Weekly Meeting Process:

For the half hour prior to start-times, the participant weighs in. Weight is recorded into a computer to track the participant's progress. The topic of the week is announced (i.e. The Sleep-Weight Loss Connection). The weekly topic is discussed amongst members and the moderator (who is a Weight Watchers lifetime member) focuses on the relationship of the topic to weight loss. All are encouraged to verbally participate but it is not a requirement. The moderator rewards members who have reached certain goals. Members also discuss their progress throughout the past week. At the end of the meeting, the moderator enforces the adoption of life-style changes to incorporate the topic of the week into daily life. Members are never pressured into buying informational products, but can do so if they decide to.

The major procedures performed for morbid obesity include the Roux-en-Y gastric bypass, sleeve gastrectomy and laparoscopic band procedure. The sleeve gastrectomy is a permanent restrictive procedure without malabsorptive components which involves a single staple line and can be performed laparoscopically in less than one hour.

While these surgical procedures are recognized as "standard" procedures for patient who have failed medical treatment and are "covered" by most health plans, access to these procedures is limited for the medically underserved, rural, poor or underrepresented minorities since national, state and municipal health plans either provide minimal coverage or no coverage at all for surgery for morbid obesity. Often, these patients wait years for elective bariatric procedures. Reimbursement to providers offering these procedures is minimal and thus access to bariatric surgery is unlikely within a timely fashion.

The laparoscopic sleeve gastrectomy involves the placement of 5 trocars. First, the V-shaped liver suspension technique (V-LIST) is used to gain a broad operative view of the gastroesophageal junction[11-12] and a silicone Penrose drain is inserted into the peritoneal cavity and stapled to the pars condensa of the lesser omentum and parietal peritoneum using 2-0 Prolene (Ethicon) for liver retraction. The left lobe of liver is retracted with the V-shaped suspension technique. The greater curvature of stomach is freed beginning from 6 cm proximal to the pylorus to the angle of His with the harmonic scalpel (Ethicon). Care is taken to preserve the gastroepiploic vessels. A bougie (36-40 Fr) is placed in the stomach against the lesser curvature to guide the stapling. Gastric resection is performed with a stapler (Echelon 60, Ethicon) along a line parallel to the bougie beginning from 6 cm proximal to the pylorus and extending to the cardia. The remnant stomach is removed from the abdominal cavity by slightly enlarging the incision where the Versaport cannula has been placed. A leak check may be performed at the same time by insufflating with a gastroscope with the remnant gastric section submerged in irrigation fluid and by infusing sterile methylene blue through a nasogastric tube. The staple line may also be oversewn (3-0 Vicryl, Ethicon), only along the bleeding and leakage areas, or areas with the potential for such complications. A nasogastric decompression tube may be placed to monitor bleeding and an intraperitoneal drain placed under an anastomotic stoma.

For the purposes of this study we will consider the following to meet the criteria of populations that are underserved, rural, poor and/or underrepresented:

Medically Underserved Populations Populations that have inadequate access to, or reduced utilization of, high-quality cancer prevention, screening and early detection, treatment, and/or rehabilitation services. Included are rural, low-literacy, and low-income populations. An effort to clarify and further define "medically underserved" is currently underway at NIH.

Rural The working definition of rural, taken from the U.S. Census Bureau, is somewhat vague. "Rural" is defined as territory, populations, and housing units not classified as "urban." The Census Bureau's definition of "urban" is places of 2,500 or more persons incorporated as cities, villages, boroughs, and towns.

Poor (Low Income)

The 1998 DHHS Poverty Guidelines (also referred to as the "Federal poverty level") define a poverty threshold as an annual income of approximately $10,000 for a single individual and an annual income of approximately $20,000 for a family of 4 (Federal Register 63, #36, February 24, 1998, pp 9235-9238).

Underrepresented Minority

For NCI purposes, a person is an underrepresented minority if he or she belongs to a minority group that is underrepresented in biomedical and behavioral science careers, based on their minority group's representation in the total population. Using this definition and available data on minority representation in the health professions, science, and engineering, blacks, Hispanics, American Indian or Alaskan Native, and Pacific Islanders are classified as underrepresented minorities. Asians are not considered to be an underrepresented minority.

The bariatric surgical procedures, including the sleeve gastrectomy, performed at UCSF by the principal investigator, Dr. Stanley J. Rogers, (Chief of Minimally Invasive Surgery and Surgical Director of Bariatric Surgery) for the past 5 years, has a documented zero percent mortality, a mean 98% laparoscopic completion rate and a mean duration of hospitalization under 3 days. The cost of these procedures also is relatively inexpensive while requiring less than 2 hours of surgery time.

We propose to randomize patients to a surgical arm (sleeve gastrectomy) plus the Weight Watchers program or to the Weight Watchers program alone. We will employ extensive metrics to assess the impact of laparoscopic sleeve gastrectomy surgery plus Weight Watchers vs. Weight Watchers Program alone monitoring for 12 months the following:

Weight reduction efficacy Self-worth assessment Health care cost Economic productivity Stress and anger Intergenerational impact

ELIGIBILITY:
Inclusion Criteria: Patients who are morbidly obese.

1. Female, age 18-65 years
2. Meeting the criteria as outlined in Part 2 A (Synopsis) of a medically underserved, rural, poor or underrepresented minority.
3. BMI > 40 and < 55, or BMI > 35 and <55 with one or more significant comorbidities. Co-morbidities are defined as diabetes, pulmonary disease, cardiac disease, or hypertension [systolic blood pressure of ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg (or both) or on treatment for hypertension]
4. History of obesity for at least 2.5 years
5. History of failure with non-surgical weight loss methods
6. Agree to comply with the substantial dietary restrictions and exercise program required by the procedure
7. Signed approval by physician and psychologist of subject's physical and mental suitability for bariatric surgery
8. Understands risks of procedures, agree to follow protocol requirements, including signing informed consent, returning for follow-up visits and completing all required testing, completing diet and behavior modification counseling.
9. Subject is a resident within the state of California or the city of Bangkok, Thailand and will likely remain so for a 2 year period of time.
10. Willingness to participate in weekly visits with Weight Watchers International local program.

Exclusion Criteria:

1. Subject history of inflammatory disease of the gastrointestinal tract including Crohn's disease or ulcerative colitis
2. Significant known esophageal disease including grade 3-4 esophagitis, active gastric ulcer disease or active duodenal ulcer disease
3. Severe coagulopathy, upper GI bleeding conditions such as esophageal or gastric varices, congenital or acquired telangiectasia
4. Congenital or acquired anomalies of the GI tract such as atresias or stenoses.
5. Severe cardiopulmonary disease or other serious organic disease including HIV or cancer
6. Currently pregnant or nursing. Potentially childbearing (i.e. not post-menopausal or surgically sterilized) and not willing to use an effective method of contraception for the next 12 months
7. Current alcohol or drug addiction
8. Mentally retarded or emotionally unstable, or exhibits psychological characteristics which, in the opinion of the investigator or psychologist/psychiatrist, make the subject a poor candidate for this procedure
9. Previous gastric, esophageal, pancreatic, or bariatric surgery
10. Infection anywhere in the body at the time of the procedure
11. Subject history of scleroderma, amyloidosis
12. Thyroid disease which is not controlled with medication
13. Hormonal or genetic cause for the obese state.
14. History of cancer other than localized basal cell carcinoma.
15. Myocardial infarction or cerebrovascular accident within past year.
16. Angina pectoris.
17. Severe coagulopathy (prothrombin time > 3 seconds over control or platelet count < 100,000)
18. Gastroparesis or pyloric stenosis.
19. Lesions with increased risk of bleeding.
20. Severe cardiopulmonary disease or other serious organic disease, including HIV or cancer.
21. Congestive heart failure.
22. Uncontrolled hypertension (systolic > 150 or diastolic > 100).
23. Severe or advanced liver disease (such as cirrhosis, chronic hepatitis, portal hypertension, etc.).
24. Severe reflux disease.
25. Active, continuous alcohol consumption (> 80 gm/day of ethanol) or chronic illicit drug use within the last 3 years.
26. Currently on prescription or over the counter diet drugs.
27. Chronic therapy with aspirin, NSAID or anticoagulants.
28. Not ambulatory.
29. Participating in another ongoing clinical trial in which concomitant diagnosis or therapeutic intervention would adversely affect the integrity of the clinical trial.

    -

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
body mass index (BMI) | One year post randomization (% of patients with reduction in BMI by 5 points)
  Comparison of body mass index (BMI) in underserved young women treated with laparoscopic sleeve gastrectomy plus Weight Watchers vs. Weight Watchers alone for the treatment of morbid obesity .

SECONDARY OUTCOMES:
quality of life | One year after study completion
  Determine the effect of treatment on quality of life, employability, income levels, overall costs to society and co-morbidities

CONTACTS AND LOCATIONS:
Overall Officials: John P Cello, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF/San Francisco General Hospital, San Francisco, California, United States